CLINICAL TRIAL: NCT07049237
Title: Effects of Evidence-Based Nursing Under a Quantitative Assessment Strategy on Cancer-Related Fatigue, Self-Management Ability, and Quality of Life in Lung Cancer Patients Undergoing Chemotherapy
Brief Title: Evidence-Based Nursing for Fatigue and Quality of Life in Lung Cancer Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Feifei Wang, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023S00501
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: Chemotherapy; Cancer-Related Fatigue; CRF; Self-Management Ability; Quality of Life; QoL; Evidence-Based Nursing; Quantitative Assessment Strategy; Edmonton Symptom Assessment Scale
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-Based Nursing Under Quantitative Assessment Strategy (EB-NQAS) Group (Experimental): Participants (n=75) received evidence-based nursing under a quantitative assessment strategy. This involved baseline assessment with ESAS; tailored care planning for pain, fatigue, nausea/vomiting, and psychological distress (including CBT, activity/sleep plans, prophylactic antiemetics); and dynamic daily/weekly evaluation and adjustment of care based on ESAS scores.
  Interventions: Behavioral: Evidence-Based Nursing Under Quantitative Assessment Strategy (EB-NQAS)
- Routine Nursing Care Group (Active Comparator): Participants (n=75) received standard nursing care as per hospital guidelines, including health education on lung cancer and chemotherapy, weekly 15-minute psychological support sessions, individualized dietary guidance, and verbal instructions on managing adverse effects.
  Interventions: Behavioral: Routine Nursing Care

INTERVENTIONS:
Behavioral: Evidence-Based Nursing Under Quantitative Assessment Strategy (EB-NQAS) — A multifaceted nursing program using the Edmonton Symptom Assessment Scale (ESAS) for quantitative symptom assessment to guide personalized, evidence-based care plans. Interventions included tailored strategies for pain management (graded, music therapy, heat, opioids), fatigue (supervised walking, sleep optimization), nausea/vomiting prevention (prophylactic antiemetics, ginger, dietary advice), and psychological support (cognitive-behavioral therapy). Care plans were dynamically monitored and adjusted.
  Arms: Evidence-Based Nursing Under Quantitative Assessment Strategy (EB-NQAS) Group
Behavioral: Routine Nursing Care — Standard hospital oncology nursing care including health education, general psychological support (weekly 15-minute sessions), dietary guidance based on nutritional risk screening, and verbal instructions for managing common adverse effects.
  Arms: Routine Nursing Care Group

SUMMARY:
This prospective randomized controlled trial investigated the effects of an evidence-based nursing intervention under a quantitative assessment strategy (EB-NQAS), utilizing the Edmonton Symptom Assessment Scale (ESAS), on cancer-related fatigue, self-management ability, and quality of life in lung cancer patients undergoing chemotherapy. Outcomes were compared to a group receiving routine nursing care.

DETAILED DESCRIPTION:
Lung cancer patients undergoing chemotherapy frequently experience significant cancer-related fatigue (CRF) and diminished quality of life (QoL), which may not be adequately addressed by conventional nursing approaches. This study aimed to evaluate the efficacy of an evidence-based nursing intervention guided by a quantitative assessment strategy (EB-NQAS). The EB-NQAS group (n=75) received personalized care plans developed by a dedicated nursing team. These plans were based on quantitative symptom assessment using the Edmonton Symptom Assessment Scale (ESAS) and incorporated evidence-based interventions for pain management (e.g., graded approach, music therapy, opioids), fatigue (e.g., activity plans, sleep optimization), nausea/vomiting prevention (e.g., prophylactic antiemetics, ginger, dietary advice), and psychological support (e.g., cognitive-behavioral therapy). Care plans were dynamically evaluated and adjusted based on daily and weekly ESAS monitoring. The control group (n=75) received routine nursing care, including standard health education, psychological support, dietary guidance, and adverse effect management. The study compared the effects of EB-NQAS versus routine nursing on CRF, self-management ability, QoL, and adverse events over a 3-month intervention period in 150 randomized lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or radiologically confirmed lung cancer (World Health Organization [WHO] 2021 diagnostic criteria).
* Scheduled to receive first-line chemotherapy (platinum-based regimen).
* Karnofsky Performance Status (KPS) score ≥60.
* Estimated survival time >6 months (assessed by treating oncologist).
* Normal mental and cognitive function (Mini-Mental State Examination [MMSE] score ≥24).
* Voluntary participation and signed informed consent.

Exclusion Criteria:

* Concurrent severe organ dysfunction (Child-Pugh score ≥B for liver; estimated glomerular filtration rate [eGFR] <30 mL/min/1.73m² for kidney).
* Active neurological disorders (e.g., stroke, epilepsy) affecting symptom reporting.
* Acute infectious diseases (e.g., tuberculosis with sputum positivity).
* Known allergies to chemotherapy drugs (e.g., platinum agents).
* Acute illnesses requiring hospitalization (e.g., pneumonia, myocardial infarction).
* Secondary malignancies (pathologically confirmed).
* Chemotherapy contraindications (e.g., uncontrolled heart failure).
* Inability to communicate in the local language (assessed via nurse interview).
* Concurrent radiotherapy or immunotherapy.
* Participation in other interventional clinical trials within 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Cancer-Related Fatigue (CRF) | Baseline, 1 month, and 3 months post-intervention.
  Assessed using the Piper Fatigue Scale (PFS). The PFS consists of 22 items covering 4 domains (behavioral, emotional, cognitive, physical), with each item scored from 0 to 10. The total score ranges from 0 to 220, where higher scores indicate more severe fatigue.

SECONDARY OUTCOMES:
Change in Self-Management Ability | Baseline, 1 month, and 3 months post-intervention.
  Evaluated using the Adult Health Self-Management Scale (AHSMSRS). This 38-item scale assesses 3 domains (environment, behavior, cognition), with items scored from 1 to 5. The total score ranges from 38 to 190, with higher scores indicating better self-management ability.
Change in Quality of Life (QoL) | Baseline, 1 month, and 3 months post-intervention.
  Measured using the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC-QLQ-C30). This questionnaire assesses 4 functioning domains and 5 symptom domains. Scores are normalized to a 0-100 scale; higher scores represent better functioning/QoL for functioning scales and more severe symptoms for symptom scales.
Incidence of Chemotherapy-Related Adverse Events | Assessed daily during the intervention period (up to 3 months).
  Occurrence of chemotherapy-related adverse effects, including gastrointestinal reactions (nausea/vomiting ≥CTCAE grade 2), hepatic dysfunction (AST/ALT >2 times Upper Limit of Normal), myelosuppression (neutrophils <1.5×10⁹/L), neurotoxicity (peripheral numbness ≥grade 2), and alopecia. Adverse events were recorded daily using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China